CLINICAL TRIAL: NCT05417906
Title: Investigating the Blood Eosinophil Count as a Biomarker to Guide Systemic Corticosteroid Treatment in Hospitalized Exacerbations of Asthma: a Randomized, Controlled, Open-label, Noninferiority Trial
Brief Title: Using the Blood Eosinophil Count to Guide Systemic Corticosteroid Treatment in Asthma Exacerbations
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Changi General Hospital (Other)
Collaborators: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03/FY2021/P2/10-A91
Record Dates: First submitted 2022-05-29; First posted 2022-06-14 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Asthma Attack; Asthma
MeSH Terms: conditions — Asthma | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard care (Active Comparator)
  Interventions: Other: Standard care
- Eosinophil-directed care (Experimental)
  Interventions: Other: Eosinophil-directed care

INTERVENTIONS:
Other: Standard care — Oral prednisolone for 5 days
  Arms: Standard care
Other: Eosinophil-directed care — Oral prednisolone for 5 days if eosinophil count is ≥ 0.300 x 10^3/µL, or 3 days if eosinophil is < 0.300 x 10^3/µL
  Arms: Eosinophil-directed care

SUMMARY:
Asthma attacks which are moderate-to-severe are typically treated with corticosteroids, but the optimal treatment duration is unknown and treatment responses can be variable. Inadequate treatment may compromise recovery, but increased exposure to corticosteroids is, in turn, associated with drug-related adverse effects.

There is a need for a biomarker to guide duration of corticosteroid treatment in asthma attacks. One such candidate biomarker is the blood eosinophil count, which may predict steroid-responsiveness. We hypothesize that the blood eosinophil count can potentially be used as a biomarker to guide the duration of corticosteroids in moderate-to-severe asthma attacks.

This study will recruit individuals hospitalized for asthma attack. Participants will be randomized to standard care or blood-eosinophil guided systemic corticosteroid therapy. Subjects in the standard arm will receive oral corticosteroids for a total of 5 days. Subjects in the blood-eosinophil guided arm will receive oral corticosteroids for a total of 5 days if admission eosinophil count is ≥ 0.300 x 10^3/µL, and receive 3 days of oral corticosteroids if the admission blood eosinophil is < 0.300 x 10^3/µL. The rate of treatment failure will be compared between these two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 21 years old
2. Admitted for acute exacerbation of asthma and have received ≤ 3 days of systemic corticosteroids
3. Have a had a blood eosinophil count (as part of routine clinical care) drawn before administration of systemic corticosteroid
4. Have not taken SCS within 7 days prior to presentation to hospital

Exclusion Criteria:

1. Concomitant pneumonia
2. Admission to high-dependency/intensive care unit, or requirement for invasive/noninvasive mechanical ventilation
3. Eosinophilia due to other known causes (eosinophilic granulomatosis and polyangiitis, parasitic infections, malignancy)
4. Other concomitant respiratory conditions e.g. chronic obstructive pulmonary disease, bronchiectasis
5. Those on anti-IL5 or anti-IL5R treatment
6. Pregnant subjects
7. Subjects who are already on an investigational drug or has been participating in another clinical study with an investigational product within the last 6 months
8. Subjects deemed by investigators to have a life expectancy of < 12 months (any cause)
9. Prisoners

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-06-02 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants experiencing treatment failure | Through the duration of the index admission for asthma attack, typically 3-5 days
  Defined as death from any cause, or need for invasive/noninvasive mechanical ventilation, or need to restart/extend systemic steroid treatment

SECONDARY OUTCOMES:
Length of hospital stay (number of days) | Through the duration of the index admission for asthma attack, typically 3-5 days
Cumulative steroid dose at index admission (mg prednisolone-equivalent) | Through the duration of the index admission for asthma attack, typically 3-5 days
Proportion of participants receiving additional systemic steroid course within 14 days | 14 days
Asthma Control Questionnaire-5 | At baseline, 7, 14, 30 and 90 days
Proportion of participants experiencing all-cause death | 30 and 90 days
Proportion of participants who develop pneumonia | 30 and 90 days
Proportion of participants who develop venous thromboembolism | 30 and 90 days
Proportion of participants who develop sepsis | 30 and 90 days
Proportion of participants who develop fractures | 30 and 90 days
Proportion of participants who develop upper gastrointestinal bleeds/peptic or gastric ulcers | 30 and 90 days
Time to next emergency department visit or admission for asthma | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Yii, MB BChir, Principal Investigator — Changi General Hospital
Locations (2):
- Singapore (2):
  - Singapore General Hospital, Singapore
  - Changi General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yii A, Tay TR, Lee KCH, Chew SY, Sieow NY, Choo XN, Toh MR, Loh SCH, Tiew PY, Koh JMK, Tee AKH, Koh MS. Blood eosinophil-guided systemic corticosteroid duration in adults hospitalised for asthma exacerbation: a randomised, controlled, open-label, non-inferiority trial. Thorax. 2025 Dec 3:thorax-2025-223961. doi: 10.1136/thorax-2025-223961. Online ahead of print. PMID 41339088